CLINICAL TRIAL: NCT00024388
Title: Phase II Open-Label Study of Taxoprexin (DHA-Paclitaxel) Injection by 2-Hour Intravenous Infusion In Patients With Metastatic, Locally Advanced, or Unresectable Renal Cell Carcinoma
Brief Title: Chemotherapy in Treating Patients With Metastatic Kidney Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Theradex (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068928; THERADEX-P01-00-07; CCF-IRB-4046; PROTARGA-P01-00-07
Record Dates: First submitted 2001-09-13; First posted 2004-01-14 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2002-06

CONDITIONS: Kidney Cancer
Keywords: stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — docosahexaenoyl-paclitaxel

INTERVENTIONS:
Drug: DHA-paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of DHA-paclitaxel in treating patients who have locally advanced, metastatic, or unresectable kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the tumor response rate, duration of response, and time to disease progression in patients with locally advanced, metastatic, or unresectable renal cell cancer treated with DHA-paclitaxel. II. Determine the overall survival of patients treated with this drug. III. Determine the toxicity profile of this drug in these patients. IV. Assess the quality of life of patients treated with this drug.

OUTLINE: This is a multicenter study. Patients receive DHA-paclitaxel IV over 2 hours on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at baseline, every 2 courses, and at completion of treatment. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 21-50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed renal cell cancer Locally advanced OR Metastatic OR Unresectable Measurable disease No known or clinical evidence of CNS metastasis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT or SGPT no greater than 2.5 times ULN Renal: Creatinine no greater than 2.5 mg/dL Cardiovascular: No uncontrolled ventricular arrhythmia No myocardial infarction within the past 3 months No superior vena cava syndrome Neurologic: No peripheral neuropathy greater than grade 1 No uncontrolled major seizure disorder No spinal cord compression Other: No other prior malignancy except: Curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix OR Cancer curatively treated with surgery alone that has not recurred for more than 5 years No concurrent serious infection requiring parenteral therapy No unstable or serious concurrent medical conditions No psychiatric disorder that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 6 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 28 days since prior immunotherapy No concurrent immunotherapy Chemotherapy: No prior chemotherapy for advanced disease No prior taxanes At least 28 days since prior chemotherapy No other concurrent chemotherapy Endocrine therapy: At least 28 days since prior hormonal therapy No concurrent hormonal therapy Radiotherapy: At least 28 days since prior large-field radiotherapy No concurrent radiotherapy Surgery: At least 14 days since prior major surgery Other: Concurrent bisphosphonates allowed if on stable dose for at least 30 days prior to study No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-04

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M. Bukowski, MD, Study Chair — The Cleveland Clinic
Locations (7):
- United States (7):
  - Arizona Oncology Associates, Tucson, Arizona
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Lucille Parker Markey Cancer Center, University of Kentucky, Lexington, Kentucky
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio